CLINICAL TRIAL: NCT04192409
Title: Glycemic Control Using Mobile-based Intervention in Patients With Diabetes Undergoing Coronary Artery Bypass to Promote Self-management
Acronym: GUIDEME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FW2019-1151
Record Dates: First submitted 2019-10-30; First posted 2019-12-10 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-06

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass; Diabetes Mellitus
Keywords: Coronary Artery Disease; Coronary Artery Bypass Grafting; Diabetes Mellitus; Smartphone Application; Postoperative Management
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-Smartphone Application (Experimental): Patients will install a smartphone application that custom-developed for the study and learn to use it with the help of researchers. The application will have the following functions: 1) providing health education information about glycemic control, postoperative management and important of drug compliance; 2) providing alert & record service on patients' DM and CAD medication treatment; 3) aiding patients to conduct self-evaluate by providing questionnaire about patients' recent basic health parameters on times. The information will be interpreted automatically by application and brief feedback will be provided to patients; 4) recording patients' fasting plasma glucose value that input by patients and generate a recent glycemic control report.
  Interventions: Behavioral: Smartphone Application
- Control (No Intervention): Patients will receive no additional intervention from researchers except the usual care provided by hospital.

INTERVENTIONS:
Behavioral: Smartphone Application — Patients will use a smartphone application contain the following functions: providing health education information about DM and CAD, reminding patients to take medicine on time by alarm, recording patients' recent fast plasma glucose value.
  Arms: Intervention-Smartphone Application

SUMMARY:
The study is a two-arm parallel, randomized clinical trial. The purpose of the study is to evaluate the effectiveness and feasibility of using high-quality medication reminder smartphone application as a tool for secondary prevention in patients undergone CABG with DM, including the change in quality of life, medication adherence improvement and clinical outcome. The participants will be randomized into intervention and control groups in a 1:1 ratio. The intervention group will receive information of secondary prevention of CHD and medication alarm using a specific smartphone application, while the control group will receive usual care.

DETAILED DESCRIPTION:
Objective: this study designed to evaluate the effectiveness and feasibility of using high-quality medication reminder smartphone application as a tool for secondary prevention in patients undergone CABG with DM, including the change in quality of life, medication adherence improvement and clinical outcome.

Study design: the study is a two-arm, parallel, randomized clinical trial. Patients will be eligible if they have undergone CABG at this admission, have a history of diabetes mellitus, have the capability of reading and using smartphone application, and are able to provide informed consent. Patients will be excluded if they do not have smartphone. The eligible participants will be allocated into intervention and control groups in a 1:1 ratio randomly. The intervention group will receive intervention of smartphone application in addition to usual care, while the control group will receive usual care. All the participants will be followed up for 6 months.

Study intervention: participants in the intervention group will install a specific costume smartphone application, which will send health education information, medication alarm and risk factor questionnaire at a fixed frequency to aid patients' self-evaluation, recording patients' recent fast plasma glucose value in addition to usual care.

Outcome measures: The primary endpoint is the change in glycemic hemoglobin (HbA1C). Secondary endpoints include MACCE, medication adherence, quality of life and status of graft vessel.

Statistical analysis: Evaluation will be carried out on an intention-to-treat basis. Values of analyzed endpoints between intervention group and control group will be compared according to the analysis plan. We'll follow a prespecified analysis plan and subgroup analysis will be conducted accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose with type 2 diabetes before this administration;
* Postoperative patients undergoing CABG in this hospitalization;

Exclusion Criteria:

* Die before discharge;
* Disability of reading, vision or hearing which leads to disability of using smartphone;
* Cognitive communication impairments or communication disorder;
* Unable to use smartphone.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1038 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in glucose level measured by HbA1C level | Baseline; 6 months
  We will measured the change in glucose level from baseline to 6 months.

SECONDARY OUTCOMES:
The incidence of all-cause death | 6 months
  We will measure the incidence of all-cause death at 6 months.
The incidence of major adverse cardiovascular events(MACE) | 6 months
  We will measure the incidence of major adverse cardiovascular events(MACE) at 6 months.
EQ-5D | 6 months
  We will measure the change in EQ-5D health survey 6 months postoperatively.
Medication adherence | 6 months
  Medication adherence is collected by a self-reported questionnaire including two questions: 1) have you ever forget to take your medication? If so, how often will you describe? 2) have you ceased to take any medication? If so, does it ceased as prescribed by doctor? Question 1 has four option if patients choose yes: 1) I hardly forget to take my medicine; 2) I forget to take my medicine monthly; 3) I forget to take my medicine every week; 4) I hardly take any medicine.
Status of the graft vessels | 6 months
  We will measure the status of the graft vessels by coronary CT angiography at 6 months.
blood pressure | 6 months
  We will document blood pressure at 6 months postoperatively.
blood glucose | 6 months
  We will document blood glucose at 6 months postoperatively.
low density lipoprotein | 6 months
  We will document low density lipoprotein at 6 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Feng, MD, PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Chinese Academy of Medical Science,Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Song Y, Nan Y, Feng W. Glycaemic control using mobile-based intervention in patients with diabetes undergoing coronary artery bypass-study protocol for a randomized controlled trial. Trials. 2023 Sep 13;24(1):585. doi: 10.1186/s13063-023-07580-x. PMID 37705074